CLINICAL TRIAL: NCT05830058
Title: Phase II Randomized Controlled Trial of Biologically Guided Stereotactic Body Radiation Therapy in Oligoprogressive Non-Small Cell Lung Cancer, Melanoma, and Renal Cell Carcinoma
Brief Title: Positron Emission Tomography (PET) Guided Stereotactic Body Radiation Therapy for the Treatment of Oligoprogressive Non-small Cell Lung Cancer, Melanoma, and Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22350; NCI-2023-02155 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22350 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-17; First posted 2023-04-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Lung Non-Small Cell Carcinoma; Malignant Solid Neoplasm; Melanoma; Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARM I: (standard care SBRT) (Experimental): Patients undergo 5 SBRT treatments every other day on study. Patients also undergo CT or PET/CT and blood collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy
- ARM II: (PET guided SBRT) (Experimental): ARM II: Patients undergo 3 SBRT treatments every other day week 1, undergo PET/CT and replanning one month post SBRT, then undergo 2 additional treatments with SIB on study. Patients also undergo CT or PET/CT and blood collection throughout study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial tests the safety of positron emission tomography (PET) guided stereotactic body radiation therapy (SBRT) and how well it works to treat non-small cell lung cancer (NSCLC), melanoma, and renal cell carcinoma (RCC) that has up to 5 sites of progression (oligoprogression) compared to standard SBRT. SBRT uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. A PET scan is an imaging test that looks at your tissues and organs using a small amount of a radioactive substance. It also checks for cancer and may help find cancer remaining in areas already treated. Using a PET scan for SBRT planning may help increase the dose of radiation given to the most resistant part of the cancer in patients with oligoprogressive NSCLC, melanoma, and RCC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. PET adaptive SBRT is both feasible and safe and allows for a higher total dose of radiation through an inter-fraction simultaneous integrated boost (SIB) based on inter-fraction PET uptake, leading to improved local control outcomes compared to current standard SBRT planning without a SIB.

SECONDARY OBJECTIVES:

I. Determine the duration of local and distant control followed PET adaptive SBRT treatment compared to standard external beam radiation therapy (EBRT).

II. Evaluate the utility of measuring circulating tumor deoxyribonucleic acid (DNA) (ctDNA) before, during and after SBRT in conjuction with biological imaging to assess early disease response.

III. Identify genomic predictors to predict for distant progression. IV. Determine durability of current systemic therapy with SBRT to oligoprogressive sites.

EXPLORATORY OBJECTIVES:

I. Biomarker changes based on ctDNA before, during and after treatment. II. Changes in fludeoxyglucose (FDG) uptake with SBRT and combined checkpoint inhibitor during and after treatment and correlation with local and distant control.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo 5 SBRT treatments every other day on study. Patients also undergo computed tomography (CT) or PET/CT and blood collection throughout study.

ARM II: Patients undergo 3 SBRT treatments every other day week 1, undergo PET/CT and replanning one month post SBRT, then undergo 2 additional treatments with SIB on study. Patients also undergo CT or PET/CT and blood collection throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: >= 18 years
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically or cytologically confirmed NSCLC with 1-5 sites of disease progression while on or following systemic therapy with a checkpoint inhibitor with or without chemotherapy for at least 3 months with radiographic evidence of progression based on Response Evaluation Criteria in Solid Tumors (RECIST) or Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST)
* Lesion(s) must all be amenable to SBRT which will be determined by the radiation oncologists. Active lesions should be a minimum size of >= 1 cm
* Primary tumor should be controlled for > 3 months in the metachronous setting; for synchronouos progression of the primary and oligoprogressive site(s), the primary should be treated with curative/local control intent
* Patients eligible for the study must have at least one lesion for which the planned radiation dose achieves a biologic effective dose (BED) < 100 (alpha/beta = 10) due to organs at risk and dose constraints
* If the clinical scenario deem that other forms of local therapy may be more suitable for the metastatic disease, such as surgical resection and interventional radiology-guided ablation, patients would be able to undergo other forms of local therapy after discussion with the study PI but at least one lesion must be treated with SBRT in this scenario
* Patients with brain metastases can be included but brain metastases must be treated prior to enrollment and are not considered as a site of oligoprogression
* Life expectancy >= 3 months in the opinion of the treating investigators

Exclusion Criteria:

* Judgement by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions, and requirements
* Those not eligible for SBRT after review by a radiation oncologist
* Unable to undergo a Pet/CT or do not have Pet active disease
* Pregnant and/or breastfeeding women are excluded from this study as these agents may have the potential for teratogenic or abortifacient effects. Female patients of childbearing potentially must have a negative urine or serum pregnancy test within 72 hours prior to receiving therapy
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2027-02-03 (Estimated); Study Completion 2027-02-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety of positron emission tomography (PET) adaptive stereotactic body radiation therapy (SBRT) | At completion of SBRT up to 5 weeks
  Feasibility and safety of biologically-guided adaptive planning based on the standardized uptake value (SUV) on pre-treatment and inter-fraction FDG-PET/CT to guide SBRT dose-escalation with a simultaneous integrated boost (SIB) delivered to areas of higher activity in patients with oligoprogressive (1-5 sites) disease when compared to the current standard SBRT planning without inter-fraction adaptive planning, with the goal of demonstrating that PET-adaptive inter-fraction planning can improve total dose delivered over the course of treatment. We will be measuring the difference in total radiation dose in Gy between the two arms with the goal of achieving an absolute dose of 10 Gy or higher.

SECONDARY OUTCOMES:
Time to progression | Up to 12 months
  Defined as time of randomization to disease progression at any site or death. Assessed using the modified Response Evaluation Criteria in Solid Tumors (mRECIST).
Time to next systemic therapy | Up to 12 months
Overall survival | Up to 12 months
Quality of life (QOL) | Up to 12 months
  Patient reported outcomes using the Functional Assessment of Cancer Therapy - G. Baseline changes in reported QOL will be summarized. Repeated QOL assessments will be tabulated and graphically displayed to describe the changes of QOL outcomes over time, no formal hypothesis testing is planned. An evaluation by dose, response and other characteristics may also be considered. For quantitative QOL scales, data will be represented using means/ medians, histogram/ boxplots. The area under curve will be used as a summary score for each patient. These can then be averaged across groups for informal assessment. Standard imputation methods will be used to deal with a large proportion of missing data.
Incidence of adverse events | At 3, 6, and 12 months following radiation therapy
  Clinician documented toxicity using common terminology for adverse events version 5.
Local control rates | Up to 12 months
  Assessed using the mRECIST.
Dose delivered | Up to 12 months
  Defined as the dose delivered in the experimental group for the first 3 fractions versus the dose given for the last 2 fractions.

CONTACTS AND LOCATIONS:
Overall Officials: Arya Amini, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States